CLINICAL TRIAL: NCT02978313
Title: Biomarker-Panel Enriched Maintenance Treatment With Cetuximab Monotherapy Versus Continuation After Induction Treatment With Chemotherapy + Cetuximab in Metastatic Colorectal Cancer (mCRC)
Brief Title: Cetuximab Monotherapy Maintenance Treatment in mCRC
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ruijin Hospital (Other)
Collaborators: Jiangsu Cancer Institute & Hospital (Other); Henan Cancer Hospital (Other Government); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, Hao Li, MD &Ph.D, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RJH-Cet-Maintenance
Record Dates: First submitted 2016-09-08; First posted 2016-11-30 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-11

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab; IFL protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cet maintenance (Experimental): Cetuximab maintenance treatment following induction treatment
  Interventions: Drug: Cetuximab
- Cet+chemo continuation (Active Comparator): Cetuximab plus continuation mFOLFOX6/FOLFIRI regimens
  Interventions: Drug: Cetuximab; Drug: mFOLFOX6; Drug: FOLFIRI

INTERVENTIONS:
Drug: Cetuximab — anti-EGFR monoclonal antibody
  Other Names: erbitux
Drug: mFOLFOX6 — Oxaliplatin+LV5FU2
  Arms: Cet+chemo continuation
Drug: FOLFIRI — Irinotecan+LV5FU2
  Arms: Cet+chemo continuation

SUMMARY:
Investigating the efficacy of Cetuximab Monotherapy versus Continuation after induction treatment with chemotherapy + Cetuximab in inoperable or irresectable and non-progressive metastatic colorectal cancer after first line induction treatment for 24 weeks with mFOLFOX6/FOLFIRI and Cetuximab treatment. Reinduction treatment will be done in case of progression.

DETAILED DESCRIPTION:
Investigating the efficacy of Cetuximab Monotherapy versus Continuation after induction treatment with chemotherapy + Cetuximab in inoperable or irresectable and non-progressive metastatic colorectal cancer after first line induction treatment for 24 weeks with mFOLFOX6/FOLFIRI and Cetuximab treatment. Reinduction treatment will be done in case of progression. This treatment is continued until progression or severe toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histological proof of colorectal cancer (in case of a single metastasis, histological or cytological proof of this lesion should be obtained);
* Distant metastases (patients with only local recurrence are not eligible);
* Unidimensionally measurable disease (> 1 cm on spiral CT scan or > 2 cm on chest X-ray; liver ultrasound is not allowed). Serum CEA may not be used as a parameter for disease evaluation;
* In case of previous radiotherapy, at least one measurable lesion should be located outside the irradiated field;
* Ongoing or planned first line treatment with 6 cycles of mFOLFOX6/FOLFIRI plus Cetuximab.

At randomisation:

* WHO performance status 0-1 (Karnofsky PS > 70%);
* Laboratory values obtained ≤ 2 weeks prior to randomisation:

  * adequate bone marrow function (Hb > 6.0 mmol/L, absolute neutrophil count > 1.5 x 109/L, platelets > 100 x 109/L),
  * renal function (serum creatinine ≤ 1.5x ULN and creatinine clearance, Cockroft formula, > 30 ml/min),
  * liver function (serum bilirubin ≤ 2 x ULN, serum transaminases ≤ 3 x ULN without presence of liver metastases or ≤ 5x ULN with presence of liver metastases);
* Negative pregnancy test in women with childbearing potential;
* Expected adequacy of follow-up;
* Institutional Review Board approval;
* Written informed consent Exclusion criteria;
* History or clinical signs/symptoms of CNS metastases;
* History of a second malignancy ≤ 5 years with the exception of adequately treated carcinoma of cervix or basal/squamous cell carcinoma of skin.

Exclusion Criteria:

* Prior adjuvant treatment for stage II/III colorectal cancer ending within 6 months before the start of induction treatment;
* Any prior adjuvant treatment after resection of distant metastases;
* Previous systemic treatment for advanced disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2016-11; Primary Completion 2019-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
PFS | 4-6 months

SECONDARY OUTCOMES:
OS | 22 months
QoL | 22 months

CONTACTS AND LOCATIONS:
Overall Officials: Yifeng Wang, MD, Principal Investigator — Ruijin Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tveit KM, Guren T, Glimelius B, Pfeiffer P, Sorbye H, Pyrhonen S, Sigurdsson F, Kure E, Ikdahl T, Skovlund E, Fokstuen T, Hansen F, Hofsli E, Birkemeyer E, Johnsson A, Starkhammar H, Yilmaz MK, Keldsen N, Erdal AB, Dajani O, Dahl O, Christoffersen T. Phase III trial of cetuximab with continuous or intermittent fluorouracil, leucovorin, and oxaliplatin (Nordic FLOX) versus FLOX alone in first-line treatment of metastatic colorectal cancer: the NORDIC-VII study. J Clin Oncol. 2012 May 20;30(15):1755-62. doi: 10.1200/JCO.2011.38.0915. Epub 2012 Apr 2. PMID 22473155
- [Background] Van Cutsem E, Kohne CH, Hitre E, Zaluski J, Chang Chien CR, Makhson A, D'Haens G, Pinter T, Lim R, Bodoky G, Roh JK, Folprecht G, Ruff P, Stroh C, Tejpar S, Schlichting M, Nippgen J, Rougier P. Cetuximab and chemotherapy as initial treatment for metastatic colorectal cancer. N Engl J Med. 2009 Apr 2;360(14):1408-17. doi: 10.1056/NEJMoa0805019. PMID 19339720